CLINICAL TRIAL: NCT04820894
Title: The Perception of Cure Among Patients With Metastatic Cancer
Brief Title: Perception of Cure Among Patients With Metastatic Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Feasibility
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19322; NCI-2021-01818 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19322 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey, medical records review): Patients complete surveys over 30 minutes about sociodemographic information and perception of immunotherapy, over 10 minutes about expectations of cure, over 10 minutes about anxiety, over 10 minutes about depression, and over 30 minutes about physical well-being. Patients' medical records are reviewed.
  Interventions: Other: Electronic Medical Record; Other: Survey Administration

INTERVENTIONS:
Other: Electronic Medical Record — Medical records are reviewed
  Other Names: Computer Based Patient Record; EMR; EMR (electronic medical record)
Other: Survey Administration — Complete surveys

SUMMARY:
This study collects information about perception of cure among patients with cancer that has spread to other places in the body (metastatic). This study aims to determine patients' perception (knowledge) before starting immunotherapy and if differences exist in understanding of treatment to stimulate or restore the ability of the body's immune (defense) system to fight infection and disease (immunotherapy) based on social and economic factors or on race/ethnicity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the proportion of patients with metastatic cancer who anticipate cure before starting immunotherapy.

SECONDARY OBJECTIVES:

I. To determine if expectations of cure are associated with quality of life and distress.

II. To determine if patients' perceptions differ by gender, age, and ethnicity.

OUTLINE:

Patients complete surveys over 30 minutes about sociodemographic information and perception of immunotherapy, over 10 minutes about expectations of cure, over 10 minutes about anxiety, over 10 minutes about depression, and over 30 minutes about physical well-being. Patients' medical records are reviewed.

ELIGIBILITY:
Eligibility Criteria:

1. Patients must be aged 18 and over
2. Patients sufficiently fluent in English
3. Patients must have a cytologically or pathologically verified diagnosis of cancer
4. Patients must have measurable metastatic disease
5. Patients must be initiating immunotherapy
6. Patients must be undergoing evaluation and treatment at City of Hope Cancer Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients | Up to 2 years
  Will assess the percentage of patients who anticipate cure before starting immunotherapy, scoring a '1' on the Perception of cure tool, and anticipate >75% chance for a cure.
Patient Reported Outcomes Measurement Information System (PROMIS) | Up to 2 years
  Descriptive analyses (e.g. frequency statistics) will be used to characterize the sample and to look at the association between Patient Reported Outcomes Measurement Information System (PROMIS) tool score with perception of cure score.
Functional Assessment of Cancer Therapy-General (FACT-G) | Up to 2 years
  Descriptive analyses (e.g. frequency statistics) will be used to characterize the sample and to look at the association between Functional Assessment of Cancer Therapy-General (FACT-G) overall score with perception of cure score.
Perceptions of cure | Up to 2 years
  Chi-square analyses will be used to examine perceptions of cure by sociodemographic characteristics:
  gender (male and female), age (< 60 and > 60), and ethnicity (white non-Hispanic, Hispanic, and other).

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Medical Center